CLINICAL TRIAL: NCT06425471
Title: A Prospective Study on the Efficacy of the Karl Storz Curved Fetoscope (11508aak) and Its Straight Version (11506akk) for In-utero Surgery
Brief Title: The Use of Karl Storz Curved Fetoscope (11508aak) and Its Straight Version (11506akk) for In-utero Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jimmy Espinoza, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-1019
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: In Utero Procedure Affecting Fetus or Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- KARL STORZ fetoscope arm (Experimental)
  Interventions: Device: KARL STORZ fetoscope arm

INTERVENTIONS:
Device: KARL STORZ fetoscope arm — The type of fetoscope used in utero(either straight or curved or both ) will depend on the location of the placenta. The fetoscope will be used to cauterize abnormal blood vessels that cause twin-to-twin transfusion syndrome (TTTS)

SUMMARY:
The purpose of this study is to prospectively evaluate the efficacy of KARL STORZ curved fetoscope (11508AAK) and its straight version (11506AAK) for in-utero surgery

DETAILED DESCRIPTION:
Outcome data will be compared to that of The Fetal Center's historical control group that underwent in-utero surgery without curved fetoscopes

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* The patient fulfills the criteria for in-utero surgery based on the standard of care, which is specific for each condition
* Patient of the baby provides signed informed consent that details the maternal and fetal risks involved with the procedure

Exclusion Criteria:

* Contraindication to abdominal surgery, fetoscopic surgery, or general anesthesia
* Allergy or previous adverse reaction to a study medication specified in this protocol
* Preterm labor, preeclampsia, or a uterine anomaly (e.g., large fibroid tumor) that is unavoidable during surgery in the index pregnancy
* Fetal aneuploidy, genomic variants of known significance if an amniocentesis has been performed, other major fetal anomalies or disorders that may impact the fetal/neonatal survival, or a known syndromic mutation
* Suspicion of a major recognized syndrome by ultrasound or MRI
* Maternal BMI >40 kg/m2
* High risk for fetal hemophilia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Gestational age at delivery in patients requiring percutaneous in-utero surgery | at time of delivery (about 10 weeks after in utero surgery)

SECONDARY OUTCOMES:
Number of successful procedures with completion of laser ablation of the abnormal vessels. | within 24 hours of in utero surgery
Improved visualization as assessed by the Likert scale | within 24 hours of in utero surgery
  This is reported categorically as strongly disagree, disagree, neither agree not disagree, agree and strongly agree. This is not a validated scale and does not have an official title. The minimum value is strongly disagree and the maximum value is strongly agree. Higher scores mean better outcomes.
Improved angle for laser visualization as assessed by the Likert scale | within 24 hours of in utero surgery
  This is reported categorically as strongly disagree, disagree, neither agree not disagree, agree and strongly agree
Improved ease of use of the new fetoscope as assessed by a questionnaire | within 24 hours of in utero surgery
  This is a 4 item questionnaire and each is scored from 1(poor) to 5(excellent) for a maximum score of 20 higher score indicating better outcome
Operative time in minutes | end of surgery ( about 1 hour form start of surgery)
  Time from from operative cannula insertion until it is removed
Number of fetuses alive prior to hospital discharge | time of discharge (about 48 hours after surgery)
Total number of maternal patients that present with short term morbidity | from end of surgery to within 10 weeks after surgery
  Short term morbidity includes but is not limited to, preterm labor, preterm premature rupture of membranes, or placental abruption
Total number of patients that have maternal and/or fetal perioperative complications | from end of surgery to within 10 weeks after surgery
The number of participants that develop twin-anemia-polycythemia sequence (TAPS) | from end of surgery to within 10 weeks after surgery
Total number of live births | from time of in utero surgery till delivery (about 10 weeks after surgery)
Total number of short-term morbidities | from time of in utero surgery till delivery (about 10 weeks after surgery)
  Short-term morbidities include, but are not limited to, premature delivery (<37 weeks), the need for extracorporeal membrane oxygenation (ECMO), neurological abnormalities found by MRI or ultrasound, gastrointestinal problems, oxygen support, infection and other problems associated with prematurity, including but not limited to, necrotizing enterocolitis, bronchopulmonary dysplasia, respiratory distress syndrome, and neonatal sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Espinoza, MD, MSc,FACOG, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No